CLINICAL TRIAL: NCT05653193
Title: Interferon-gamma as Adjunctive Therapy in Chronic Pulmonary Aspergillosis: a Randomised Feasibility Study
Acronym: INCAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B01674
Record Dates: First submitted 2022-11-29; First posted 2022-12-16 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pulmonary Aspergillosis; Aspergillosis
Keywords: immunotherapy; interferon gamma
MeSH Terms: conditions — Aspergillosis | interventions — interferon gamma-1b; Injections; Antifungal Agents; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antifungal (Active Comparator): Any oral triazole antifungal as per routine care
  Interventions: Drug: Antifungals as standard of care
- Antifungal plus inteferon gamma (Experimental): Any oral triazole antifungal as per routine care plus interferon-gamma three times weekly subcutaneously 50 micrograms/m2 for 3 months
  Interventions: Drug: Interferon Gamma-1B 0.1 MG Per 0.5 ML Injection PLUS antifungals as standard of care

INTERVENTIONS:
Drug: Interferon Gamma-1B 0.1 MG Per 0.5 ML Injection PLUS antifungals as standard of care — Patients starting oral antifungal treatment for chronic pulmonary aspergillosis will be randomised 1:1 to additional interferon-gamma for 3 months or no additional treatment.
  Arms: Antifungal plus inteferon gamma
Drug: Antifungals as standard of care — Patients starting oral antifungal treatment for chronic pulmonary aspergillosis will be randomised 1:1 to additional interferon-gamma for 3 months or no additional treatment.
  Arms: Antifungal

SUMMARY:
This study explores the role of treatment with interferon-gamma to improve outcomes in chronic pulmonary aspergillosis (CPA). CPA is a progressive infection caused by the fungus Aspergillus affecting patients with chronic lung disease like Chronic Obstructive Lung Disease (COPD) or previously treated tuberculosis (TB). It causes gradual destruction of lung tissue by slowly enlarging cavities, frequent secondary infections and poor quality of life. Because of its indolent nature and nonspecific x-ray findings, it often remains unrecognised for years. Around 3600 people live with CPA in the United Kingdom. Mortality from CPA may be up to 40% in five years.

Treatment for CPA relies on antifungals for prolonged periods, but only around 60% of patients improve. It is often long-term or lifelong as the response is slow and some patients experience relapses. In addition, only one class of oral antifungal drugs is licensed for CPA, and they are associated with side effects and high cost. Better treatments are needed for CPA. We do not know why many patients do not respond to treatment. Maybe CPA patients have a weakened immune system and are more susceptible to Aspergillus. Our data suggest that CPA patients produce lower amounts of ΙFNγ, a substance that facilitates the immune system's response against Aspergillus. We have also shown that, when given to patients with CPA who have failed to improve on antifungal treatment, interferon-gamma leads to improvement in important patient-centred outcomes like flares of lung disease or hospital admissions. Interferon-gamma is already in use in the National Health Service of the United Kingdom for other indications. Therefore, its use in CPA should be explored. However, CPA is a rare condition and the tolerability of interferon-gamma is not fully established in these patients. To understand whether a large-scale study is feasible in CPA, we first need preliminary data in smaller numbers of patients.

We are conducting a randomised trial of interferon-gamma in addition to antifungals in CPA. Patients with CPA starting antifungal treatment are eligible. Participants (25 per group) are randomly assigned to interferon-gamma for 12 weeks (in addition to antifungals) or antifungals only. To test whether the treatment works, we will use measurements of the cavities on chest CT scan and scores on a quality-of-life questionnaire. We will assess for tolerability of treatment at intervals similar to clinical practice. Criteria for progression to the large-scale study will be set based on the proportion of patients willing to participate, and on the proportion who complete the treatment. Data collected on those parameters will allow us to determine the number needed for a definite study.

If the large-scale study confirms our observations that interferon-gamma improves outcomes in CPA, then treatment duration can be shortened and relapses avoided. In addition, interferon-gamma can then be explored in other chronic lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CPA
* Started antifungal treatment for CPA within the last 8 weeks and received no antifungals for CPA in the 8 weeks prior
* Chest CT scan available within the 6 months prior to enrolment
* Individuals of child bearing potential agree to have pregnancy test an use highly effective contraception

Exclusion Criteria:

* Moderate to severe liver dysfunction (Child-Pugh Class B or C)
* Renal failure (eGFR <30 mL/min)
* Clinically diagnosed active depression
* Active tuberculosis or non-tuberculous mycobacterial (NTM) lung disease
* Acute infection or other event within the preceding 4 weeks which, as assessed by the investigators, might interfere with the assessment of response to treatment
* Use of any interferon formulation within the preceding six months
* Active viral hepatitis infection
* Pregnancy or breastfeeding
* Immunosuppression (>15mg prednisolone/day for at least four weeks or equivalent) within the preceding six months
* Inability to self-administer subcutaneous medications AND lack of a carer who can administer
* Participants lacking capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants retained in the intervention arm | 6 months
Proportion of target sample achieved | 3 years
Change in maximum cavity wall thickness on CT scan | 6 months

SECONDARY OUTCOMES:
Change in St George's Respiratory Questionnaire (SGRQ) score | 3 and 6 months
  The SGRQ ranges from 0-100 with higher scores indicating worse quality of life
Number of exacerbations requiring antibiotics or steroids in the six months before and after starting treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chris Kosmidis, MD, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No